CLINICAL TRIAL: NCT00068978
Title: Flow Cytometry Study of T Cell Responses to HIV Vaccines
Brief Title: Analysis of Immune Responses to HIV Vaccines
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 5R01AI047062-03 (NIH); 5R01AI047062-03 (NIH)
Record Dates: First submitted 2003-09-12; First posted 2003-09-16 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-08

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This study will evaluate a test designed to measure immune system responses to HIV and HIV vaccines.

DETAILED DESCRIPTION:
Assays for HIV-specific human CD4 and CD8 T cell immunity are needed in order to evaluate the immune response to HIV vaccines. Such assays should be robust, reproducible, and amenable to high throughput analysis of clinical specimens. Cytokine flow cytometry (CFC) assays can reliably and specifically detect human CD4 and CD8 T cell responses to AIDS-related opportunistic infections, including those caused by cytomegalovirus, Mycobacterium tuberculosis, the Mycobacterium avium complex, cryptococcus, and human papillomavirus. The purpose of this study is to devise and evaluate a similar CFC assay for the detection and quantitation of CD4 and CD8 T cell responses against HIV.

This study will evaluate a "Gag-IFNg CFC" assay by comparing the results of this assay with results from other assays of immune phenotype and function in long-term nonprogressors, untreated patients with progressive HIV disease, and recipients of candidate HIV vaccines. The study will also examine HIV-specific immune responses in HIV infected individuals who appear to exhibit significant immune protection from HIV disease.

Participants in this study will be drawn from other studies currently underway. As a part of those studies, participants will have regular blood tests. Blood samples from those studies will be used in this study. No participants will be directly enrolled in this study.

ELIGIBILITY:
Blood samples from 5 cohorts of HIV infected individuals and 2 cohorts of HIV uninfected individuals will be evaluated.

Varying stages of HIV disease are represented in these cohorts, including:

* Individuals who have been exposed but who have not seroconverted
* Individuals who have recently seroconverted
* HAART-treated patients who receive immune modulators such as IL-2 and therapeutic immunization
* HAART-treated patients who undergo structured treatment interruptions
* HAART-treated patients who have durable suppression of viremia
* HAART-treated patients who experience incomplete suppression of viremia
* HAART-treated patients followed with careful drug adherence monitoring
* Long-term nonprogressors
* Untreated progressors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. McCune, MD, PhD, Principal Investigator — University of California at San Francisco
Locations (1):
- Core Immunology Laboratory, San Francisco, California, United States

REFERENCES:
- [Result] Jacobson MA, Schrier R, McCune JM, Torriani FJ, Holland GN, O'Donnell JJ, Freeman WR, Bredt BM. Cytomegalovirus (CMV)-specific CD4+ T lymphocyte immune function in long-term survivors of AIDS-related CMV end-organ disease who are receiving potent antiretroviral therapy. J Infect Dis. 2001 May 1;183(9):1399-404. doi: 10.1086/319854. Epub 2001 Mar 30. PMID 11294673
- [Result] Aberg JA, Price RW, Heeren DM, Bredt B. A pilot study of the discontinuation of antifungal therapy for disseminated cryptococcal disease in patients with acquired immunodeficiency syndrome, following immunologic response to antiretroviral therapy. J Infect Dis. 2002 Apr 15;185(8):1179-82. doi: 10.1086/339680. Epub 2002 Apr 1. PMID 11930330
- [Result] Bredt BM, Higuera-Alhino D, Shade SB, Hebert SJ, McCune JM, Abrams DI. Short-term effects of cannabinoids on immune phenotype and function in HIV-1-infected patients. J Clin Pharmacol. 2002 Nov;42(S1):82S-89S. doi: 10.1002/j.1552-4604.2002.tb06007.x. PMID 12412840
- [Result] Jacobson MA, Bredt BM. Association of cytomegalovirus (CMV)-specific CD4+ T lymphocyte reactivity and protective immunity against acquired immunodeficiency syndrome-related CMV retinitis. J Infect Dis. 2002 Dec 1;186(11):1701-2; author reply 1702-3. doi: 10.1086/345369. No abstract available. PMID 12447752
- [Result] Hunt PW, Martin JN, Sinclair E, Bredt B, Hagos E, Lampiris H, Deeks SG. T cell activation is associated with lower CD4+ T cell gains in human immunodeficiency virus-infected patients with sustained viral suppression during antiretroviral therapy. J Infect Dis. 2003 May 15;187(10):1534-43. doi: 10.1086/374786. Epub 2003 Apr 23. PMID 12721933
- [Result] Abrams DI, Hilton JF, Leiser RJ, Shade SB, Elbeik TA, Aweeka FT, Benowitz NL, Bredt BM, Kosel B, Aberg JA, Deeks SG, Mitchell TF, Mulligan K, Bacchetti P, McCune JM, Schambelan M. Short-term effects of cannabinoids in patients with HIV-1 infection: a randomized, placebo-controlled clinical trial. Ann Intern Med. 2003 Aug 19;139(4):258-66. doi: 10.7326/0003-4819-139-4-200308190-00008. PMID 12965981
- [Result] Suni MA, Dunn HS, Orr PL, de Laat R, Sinclair E, Ghanekar SA, Bredt BM, Dunne JF, Maino VC, Maecker HT. Performance of plate-based cytokine flow cytometry with automated data analysis. BMC Immunol. 2003 Sep 2;4:9. doi: 10.1186/1471-2172-4-9. Epub 2003 Sep 2. PMID 12952557
- [Result] Karlsson AC, Martin JN, Younger SR, Bredt BM, Epling L, Ronquillo R, Varma A, Deeks SG, McCune JM, Nixon DF, Sinclair E. Comparison of the ELISPOT and cytokine flow cytometry assays for the enumeration of antigen-specific T cells. J Immunol Methods. 2003 Dec;283(1-2):141-53. doi: 10.1016/j.jim.2003.09.001. PMID 14659906
- [Result] Deeks SG, Martin JN, Sinclair E, Harris J, Neilands TB, Maecker HT, Hagos E, Wrin T, Petropoulos CJ, Bredt B, McCune JM. Strong cell-mediated immune responses are associated with the maintenance of low-level viremia in antiretroviral-treated individuals with drug-resistant human immunodeficiency virus type 1. J Infect Dis. 2004 Jan 15;189(2):312-21. doi: 10.1086/380098. Epub 2004 Jan 7. PMID 14722897
- [Result] Jacobson MA, Maecker HT, Orr PL, D'Amico R, Van Natta M, Li XD, Pollard RB, Bredt BM; Adult AIDS Clinical Trials Group and the Studies of Ocular Complications of AIDS Research Group. Results of a cytomegalovirus (CMV)-specific CD8+/interferon- gamma+ cytokine flow cytometry assay correlate with clinical evidence of protective immunity in patients with AIDS with CMV retinitis. J Infect Dis. 2004 Apr 15;189(8):1362-73. doi: 10.1086/382964. Epub 2004 Mar 31. PMID 15073672
- [Result] Karlsson AC, Younger SR, Martin JN, Grossman Z, Sinclair E, Hunt PW, Hagos E, Nixon DF, Deeks SG. Immunologic and virologic evolution during periods of intermittent and persistent low-level viremia. AIDS. 2004 Apr 30;18(7):981-9. doi: 10.1097/00002030-200404300-00005. PMID 15096800
- [Result] Sinclair E, Black D, Epling CL, Carvidi A, Josefowicz SZ, Bredt BM, Jacobson MA. CMV antigen-specific CD4+ and CD8+ T cell IFNgamma expression and proliferation responses in healthy CMV-seropositive individuals. Viral Immunol. 2004;17(3):445-54. doi: 10.1089/vim.2004.17.445. PMID 15357911
- [Result] Neuenburg JK, Sinclair E, Nilsson A, Kreis C, Bacchetti P, Price RW, Grant RM. HIV-producing T cells in cerebrospinal fluid. J Acquir Immune Defic Syndr. 2004 Oct 1;37(2):1237-44. doi: 10.1097/01.qai.0000136733.09275.fa. PMID 15385730
- [Result] Maecker HT, Rinfret A, D'Souza P, Darden J, Roig E, Landry C, Hayes P, Birungi J, Anzala O, Garcia M, Harari A, Frank I, Baydo R, Baker M, Holbrook J, Ottinger J, Lamoreaux L, Epling CL, Sinclair E, Suni MA, Punt K, Calarota S, El-Bahi S, Alter G, Maila H, Kuta E, Cox J, Gray C, Altfeld M, Nougarede N, Boyer J, Tussey L, Tobery T, Bredt B, Roederer M, Koup R, Maino VC, Weinhold K, Pantaleo G, Gilmour J, Horton H, Sekaly RP. Standardization of cytokine flow cytometry assays. BMC Immunol. 2005 Jun 24;6:13. doi: 10.1186/1471-2172-6-13. PMID 15978127
- [Result] Emu B, Sinclair E, Favre D, Moretto WJ, Hsue P, Hoh R, Martin JN, Nixon DF, McCune JM, Deeks SG. Phenotypic, functional, and kinetic parameters associated with apparent T-cell control of human immunodeficiency virus replication in individuals with and without antiretroviral treatment. J Virol. 2005 Nov;79(22):14169-78. doi: 10.1128/JVI.79.22.14169-14178.2005. PMID 16254352
- [Result] Jacobson MA, Sinclair E, Bredt B, Agrillo L, Black D, Epling CL, Carvidi A, Ho T, Bains R, Adler SP. Antigen-specific T cell responses induced by Towne cytomegalovirus (CMV) vaccine in CMV-seronegative vaccine recipients. J Clin Virol. 2006 Mar;35(3):332-7. doi: 10.1016/j.jcv.2005.09.019. Epub 2006 Jan 18. PMID 16387547